CLINICAL TRIAL: NCT05654714
Title: ModPG3 Adult and Pediatric AAMI (Association for the Advancement of Medical Instrumentation) 2018 ISO Clinical Investigation Protocol of SureBP and StepBP Algorithms
Brief Title: ModPG3 Adult/Ped ISO 81060-2:2018 Study Protocol
Status: Terminated | Type: Interventional
Why Stopped: This study was terminated early due to errors in the Algorithm, which may have an impact on the data.
Sponsor: Welch Allyn (Industry)
Responsible Party: Sponsor
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 60115909
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Blood pressure readings (Experimental): The study will be conducted in 2 parts.
  * Part 1 will test subjects using the ModPG3 Investigational device with the SureBP algorithm enabled.
  * Part 2 will test subjects using the ModPG3 Investigational device with the StepBP algorithm enabled.
  The study requires three observers. The first two observers take auscultatory readings that are averaged to use as reference blood pressures. The third observer operates the ModPG3 investigational device and records the readings for that device.
  The two clinicians taking reference readings will be blinded to each other's readings and to the investigational device readings.
  Interventions: Device: ModPG3 Investigational Device; Device: Auscultatory Equipment

INTERVENTIONS:
Device: ModPG3 Investigational Device — * Connex Vital Sign Monitor with ModPG3
  * Laptop
  * Blood Pressure Data Collection Software (not used for test report analysis)
  * USB cable
  * Power strip
  * Welch Allyn FlexiPort Reusable Blood Pressure Cuffs
Device: Auscultatory Equipment — * Reference Sphygmomanometer1
  * Reference Cuffs2
  * Dual Auscultatory Stethoscope
  * Tape measure
  * Stopwatch

SUMMARY:
Automated blood pressure cuff measurements taken by an "oscillometric device" is the standard in numerous medical settings today.

Studies show that oscillometric devices using algorithms are more accurate and consistent than devices using other non-invasive measuring techniques, especially in critical cases.

SureBP algorithm estimates BP during cuff inflation; the second, StepBP algorithm does so during deflation.

The purpose of this study is to test the algorithms contained in the ModPG3 on Adult and Pediatric subjects to determine if they meet the requirements of ISO 81060-2:2018/Amd 1:2020 Non-invasive sphygmomanometers - Part 2: Clinical investigation of intermittent automated measurement type

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to provide an informed consent or have legally authorized representative consent to participate.
* Subject must be willing and able to comply with the study procedures.
* Subject must be ≥ 3 years of age
* Subjects that are between 7 and 17 years of age must provide assent to participate in the study.
* Subject or legally authorized representative must be able to read, write, speak in English, French or Italian.
* Subjects must have an arm circumference in the range of 12-55 cm and fit into the usable range for the reference cuffs.
* Subject must be able to have blood pressures measured on the Left arm.

Exclusion Criteria:

* Lack of Informed consent.
* Subjects with deformities or abnormalities that may prevent proper application of the device under test.
* Subject is evaluated by the investigator or clinician and found to be medically unsuitable for participation in this study.
* Subjects with known heart dysrhythmias.
* The subject is in acute distress, i.e., severe pain or, severe emotional distress or agitation that would inhibit him/her from participating in the study.
* The subject has any known contraindication to blood pressure measurement.
* Subjects with compromised circulation or peripheral vascular disease.
* Subjects with clotting disorders or taking prescribed blood thinners.
* Subjects that cannot tolerate sitting for up to 1 hour.
* Subject with a blood pressure demographic that has already been filled.
* Subjects with a severe contact allergy to cuff material.
* Subjects with a history of skin fragility or breakdown, such as ecchymosis or lacerations, affecting the upper extremities that would affect the application of noninvasive blood pressure cuff.
* Subjects whose arm circumference does not fall within the unusable range for the reference cuffs.
* Subjects with no audible K5 sound.
* Subject is pregnant and/or breastfeeding.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baxter Investigational Site, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Sharing of Clinical Trial Data: Baxter is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, Baxter will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP's)
Supporting Information: Study Protocol, SAP
Time Frame: Upon approval of a legitimate research request.
Access Criteria: Research requests will be reviewed by qualified medical and scientific experts within the company. If Baxter agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of Baxter prior to the release of any data.
URL: https://www.baxter.com/clinical-trial-transparency-and-data-sharing-policy

RESULTS

PARTICIPANT FLOW:
Groups:
- Blood Pressure Readings: The study will be conducted in 2 parts.
  * Part 1 will test subjects using the ModPG3 Investigational device with the SureBP algorithm enabled.
  * Part 2 will test subjects using the ModPG3 Investigational device with the StepBP algorithm enabled.
  The study requires three observers. The first two observers take auscultatory readings that are averaged to use as reference blood pressures. The third observer operates the ModPG3 investigational device and records the readings for that device.
  The two clinicians taking reference readings will be blinded to each other's readings and to the investigational device readings.
  ModPG3 Investigational Device: • Connex Vital Sign Monitor with ModPG3
  * Laptop
  * Blood Pressure Data Collection Software (not used for test report analysis)
  * USB cable
  * Power strip
  * Welch Allyn FlexiPort Reusable Blood Pressure Cuffs
  Auscultatory Equipment: • Reference Sphygmomanometer1
  * Reference Cuffs2
  * Dual Auscultatory Stethoscope
  * Tape measure
  * Stopwatch
Period: Overall Study
Arm/Group | Blood Pressure Readings
Started | 152 (Due to early termination of the study, efficacy analysis was not completed, thus no scientific conclusions can be drawn from this study.)
Completed | 134 (Due to early termination of the study, efficacy analysis was not completed, thus no scientific conclusions can be drawn from this study.)
Not Completed | 18

BASELINE CHARACTERISTICS:
Population: Due to early termination of the study, efficacy analysis was not completed, thus no scientific conclusions can be drawn from this study.
Arm/Group | Blood Pressure Readings
Number analyzed (Participants) | 152
Age, Customized [Count of Participants; unit: Participants]
  3 - 17 years | 57
  >= 18 years | 95
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 88
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 152
Arm Circumference of ≥12-55 cm [Count of Participants; unit: Participants] — This measure reports the count of participants whose arm circumference fell within the usable range (12-55 cm).
  Participants | 152

OUTCOME MEASURES:

1. Primary Outcome: Compliance of the ModPG3 Blood Pressure (BP) Readings With ISO Requirements
Description: BP readings for all subjects will be calculated separately for systolic and diastolic blood pressure. At least three paired blood pressure values shall be taken for each subject. ISO 81060-2:2018/Amd 1:2020 Non-invasive sphygmomanometers - Part 2: Clinical investigation of intermittent automated measurement type
Time Frame: Day 1 (up to 1 hour)
Population: The study was terminated due to errors in the algorithm planned for data processing and analysis. A validated post processing algorithm for the raw data files was never finalized, so no blood pressure measurements needed for analysis are available. There is no data available to populate the outcome measure.
Groups:
- Blood Pressure Readings: Due to early termination of the study, efficacy analysis was not completed, thus no scientific conclusions can be drawn from this study
Arm/Group | Blood Pressure Readings
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to approximately 1 hour after consent; no follow-up was required.
Arm/Group | Blood Pressure Readings
All-Cause Mortality (participants affected / at risk) | 0/152
Serious Adverse Events (participants affected / at risk) | 0/152
Other Adverse Events (participants affected / at risk) | 0/152

LIMITATIONS AND CAVEATS:
This study was terminated early due to errors in the StepBP Algorithm 9104.16 and SureBP Algorithm 9305.10 from data gathered outside this study. The sponsor made the decision to update the software, which may have an impact on the data.

Due to early termination of the study, efficacy analysis was not completed, thus no scientific conclusions can be drawn from this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT05654714/Prot_002.pdf
  • Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT05654714/SAP_001.pdf